CLINICAL TRIAL: NCT06931756
Title: Effects of Uremia on Brachial Plexus Electrophysiology and Brachial Plexus Block: One Prospective Parallel Cohort Study
Brief Title: Effects of Uremia on Brachial Plexus Electrophysiology and Brachial Plexus Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20250123-09
Record Dates: First submitted 2025-03-30; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Electrical Stimulation of Nerves Produces Muscle Reflexes
Keywords: Neuron; Muscle movement; Electrical Stimulation; Electric current

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uremia group (U group) (Experimental): 1. Patients aged 18 years and above, ASA classification I-IV, BMI 18.5-29.9, planning to undergo forearm or hand surgery.
  2. Diagnostic criteria: Patients who meet the internationally recognized diagnostic criteria for uremia and require hemodialysis.
  3. Informed consent: Patients or their legal representatives must sign an informed consent form, agreeing to participate in this study and undergo related examinations and treatments.
  Interventions: Device: Neural Stimulator
- Non-uremia group (Group N) (Experimental): 1. According to the Propensity Score Matching (PSM) design for the control group, select patients aged 18 years or older, ASA classification I to IV, matched with patients in the U group in terms of age, gender, and BMI within the corresponding group, who are planned to undergo forearm or hand surgery. In addition to possibly having diabetes, patients should not have any other diseases that could cause peripheral neuropathy.
  2. Informed consent: Similar to the uremic patient group, an informed consent form must be signed.
  Interventions: Device: Neural Stimulator

INTERVENTIONS:
Device: Neural Stimulator — Adjust the neural stimulator, with a stimulation duration of 0.1 ms, a stimulation frequency of 1Hz, and a stimulation current of 1.0mA. Under ultrasound guidance, the needle tip is used to touch the radial nerve, ulnar nerve, median nerve, and musculocutaneous nerve respectively, until a clear motor response is observed in the corresponding muscles. Thereafter, the minimum stimulation threshold current is verified by reducing the current until the distal motor response disappears. If no motor response is elicited, the current intensity is appropriately increased to achieve a motor response of the extensor tendon of the radial nerve, and the flexor tendon motor responses of the ulnar nerve, median nerve, and musculocutaneous nerve.

SUMMARY:
As a late stage of renal failure, uremia not only leads to severe impairment of renal function in patients, but also often leads to a variety of complications, among which multiple peripheral neuropathy is particularly common. This lesion is mainly caused by the combination of multiple mechanisms, such as the accumulation of uremic toxins, electrolyte disorder, nutrient deficiency and factors related to hemodialysis. Therefore, it is important clinical significance to deeply explore the effects of uremia on electrophysiological properties and nerve block of brachial plexus.

At present, there are relatively few studies on the effects of uremia on the brachial plexus, especially the prospective parallel cohort studies on its electrophysiological properties and nerve block. As a new anesthetic technique, ultrasound-guided axillary brachial plexus block has the advantages of precise positioning, scientific administration, reducing complications and improved safety, but the application effect and safety in uremic patients still need to be further verified.

ELIGIBILITY:
Inclusion Criteria:

* Uremia group [group U]

  1. Patients aged 18 years and older
  2. ASA classification I-IV
  3. BMI 18.5-29.9
  4. Patients with uremia planning to undergo forearm or hand surgery
  5. Diagnostic criteria: Patients must meet the internationally recognized diagnostic criteria for uremia and require hemodialysis
  6. Informed consent: Patients or their legal representatives must sign an informed consent form, agreeing to participate in this study and undergo related examinations and treatments
* Non-uremia group [Group N]

  1. Patients aged 18 years and older
  2. ASA classification I-IV
  3. BMI 18.5-29.9
  4. Patients planning to undergo forearm or hand surgery
  5. In addition to possibly having diabetes, patients should not have any other diseases that could cause peripheral neuropathy
  6. The patient or their legal representative must sign an informed consent form, agreeing to participate in this study and receive the relevant examinations and treatments

Exclusion Criteria:

* Individuals allergic to study medications (such as ropivacaine)
* Those with contraindications to local anesthesia or nerve blockades, such as coagulation disorders, infections, etc.
* Those with severe cardiovascular or respiratory diseases
* Those unable to comply with study requirements, such as cognitive impairment, mental disorders, etc.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the minimum excitatory threshold current for motor electrical stimulation of the radial, ulnar, median, and musculocutaneous nerves between patients with uremia and those without uremia. | one year
  Under ultrasound guidance, using a high-frequency linear array transducer and a dedicated nerve stimulation needle, the nerves are localized in-plane technique under direct visualization. Adjust the nerve stimulator with a stimulation duration of 0.1 ms, a stimulation frequency of 1Hz, and a stimulation current of 1.0mA. Under ultrasound guidance, the needle tip is used to touch the radial nerve, ulnar nerve, median nerve, and musculocutaneous nerve respectively, until a clear motor response is observed in the corresponding muscles. Thereafter, the minimum stimulation threshold current is verified by reducing the current until the distal motor response disappears. If no motor response is elicited, the current intensity is appropriately increased to achieve motor responses of the extensor tendon of the radial nerve, and the flexor tendons of the ulnar nerve, median nerve, and musculocutaneous nerve.

SECONDARY OUTCOMES:
The onset time of forearm sensory block in two groups of patients | one year
  Testing the time for cold sensation disappearance using alcohol swabs
Onset time of forearm motor block in two groups of patients | one year
  Time when forearm muscle strength drops to grade 0.
The recovery time of forearm sensation in two groups of patients | one year
  Forearm tactile recovery time
Recovery time for forearm movement in two groups of patients | one year
  Time for forearm muscle strength to recover to pre-surgery status